CLINICAL TRIAL: NCT04865081
Title: First Randomised Controlled Clinical Evaluation of the Impact of Anti-Aerosol VACCIN Box on the Videolaryngoscopic Intubation Procedure
Brief Title: Clinical Evaluation of an Aerosol Protective Intubation Device on Videolaryngoscopic Intubation Difficulty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Responsible Party: Principal Investigator, Issam TANOUBI, MD, MA(ed), Associate Professor, Maisonneuve-Rosemont Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20212465
Record Dates: First submitted 2021-04-21; First posted 2021-04-29 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Intubation
Keywords: videolaryngoscopy; intubation box; aerosol box; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VACCIN box group (Experimental): The anesthesiologist will intubate the participants in the VACCIN box group while using the VACCIN box that will be placed over the participants' head.
  Interventions: Device: VACCIN box
- Control group (No Intervention): Enrolled participants in the control group will be intubated without the use of the VACCIN intubation box (standard anesthesia).

INTERVENTIONS:
Device: VACCIN box — The VACCIN box is a translucid box that can be placed over the patient's head. It has entry holes on the front and the side of the box in which nitrile gloves can be attached. The anesthesiologist can intubate with arms and hands inside the box. Its also has the capacity to create a negative pressure environment inside the box by connecting an air suction cable from the box to the OR medical aspiration line.
  Arms: VACCIN box group

SUMMARY:
The VACCIN box, an anti-aerosol intubation box for potential use on COVID-19 (SARS-CoV-2) positive patients, was designed in order to reduce the transmission risk to healthcare workers. This study will compare the safety and the ease of use of the VACCIN box to a standard intubation in healthy participants undergoing elective surgery. It is expected that intubation times and success rate of intubation in the same circumstances will be similar with and without the use of the VACCIN box.

DETAILED DESCRIPTION:
Novel ways to protect healthcare workers were developed around the world in the setting of the COVID-19 (SARS-CoV-2) pandemic. Shortage of personal protective equipment (PPE) and concern of potential viral transmission during aerosol generating procedures such as endotracheal intubation fueled the emergence of intubation boxes. However, a lack of details about their safety and efficiency remains.

This study will evaluate safety and ease of use of the VACCIN box in participants undergoing elective surgery requiring endotracheal intubation. The study design is a prospective randomized single center clinical trial comparing intubation with and without its use. It is expected that intubation times and success rate of intubation in the same circumstances will be similar with and without the use of the VACCIN box. Eligible participants will be randomized in a 1:1 ratio after informed consent.

Participants in both groups will be intubated in the same circumstances. The procedure include a midazolam anxiolysis, a rapid sequence induction without cricoid pressure of predefined dosing of remifentanil, propofol and rocuronium and monitoring of an adequate muscles paralysis and dept of anesthesia.

Anesthesiologists will intubate in both groups using specific material: McGRATH videolaryngoscope with X-Blade, 8 mm endotracheal tube (ETT) for men or 7 mm for women and the Glidescope videolaryngoscope stylet inside the ETT.

The experimental group will differ from the control group by application of the VACCIN box over the participant's head through which the anesthesiologist will intubate. Proper installation and removal of the VACCIN box will also be evaluated.

Intubations will only be done by anesthesiologists to assure patient safety. Each anesthesiologist will be assigned a practice session using the VACCIN box on an intubation mannequin prior to the study.

Time measurements throughout the procedure will be taken to obtain the outcomes measures. Vital signs, TOF, NOL index and BISpectral index monitoring are part of the protocol in order to assure an adequate anesthesia induction prior and after intubation.

A total of 60 participants will be enrolled in the study (30 in each group). Sample size calculation was based on local intubation mean time with COVID-19 pandemic protocols of 45 seconds with a 15 seconds standard deviation (SD). 26 participants per group are needed considering that an intubation time that is 30% or more over the current mean would imply that the VACCIN Box slowed down the intubation with an assumed SD of 15 seconds, a significance level of 5% and power of 90%. Sample size per group was rounded up to 30 in order to overcome possible exclusion or loss.

The primary outcome, the intubation time in seconds, will be tested for normal distribution with a D'Agostino-Pearson omnibus normality test and analyzed using a Two-tailed Student t test for unpaired groups. The intubation time will be presented as mean and standard deviation [SD].

For the secondary outcomes, the χ2 test will be used for the comparisons of the success rate of intubation at first laryngoscopy. The Mann-Whitney U test will be used to compare the ease of intubation.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery requiring general anesthesia with tracheal intubation
* ASA status I, II or III
* Good understanding of English or French

Exclusion Criteria:

* Known difficult airway
* Anticipated difficult airway (Mallampati ≥ 3, oral opening < 2.5 cm, thyromental distance < 6 cm, limited cervical mobility, significant abnormality of the upper respiratory tract, history of major surgery on airway or cervical area)
* COVID-19 positive or unknown status
* Rapid sequence contraindication
* Presence of antibiotic-resistant bacteria requiring a form of additional protective equipment
* Claustrophobia
* Chronic anxiety
* BMI ≥ 35
* Allergy or intolerance to any of the study drugs
* Emergent surgery
* Pregnancy
* Preoperative hemodynamic disturbance
* Patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-04-19 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Intubation time | Intubation time will correspond to the time interval in seconds between the preoxygenation face mask removal and the detection of end-tidal CO2 on the anesthesia monitor
  Seconds

SECONDARY OUTCOMES:
Success rate of intubation at first laryngoscopy | Immediately after the intubation
  Percentage
Ease of tracheal intubation | Immediately after the intubation
  Numeric scale of 0 to 10
VACCIN box installation time | The VACCIN box installation time will correspond to the time interval in the experimental group between the start of the VACCIN box placement over the participant's head to the removal of the preoxygenation mask before intubation.
  Seconds
VACCIN box removal time | The VACCIN box removal time will correspond to the time interval in the experimental group between the initial detection of end-tidal CO2 on the anesthesia monitor to the complete removal of the VACCIN box.
  Seconds
Breach of air tightness | Immediately after the intubation
  Percentage
Qualitative reviews on intubation with the VACCIN box | Immediately after the intubation
  Qualitative
Non-invasive blood pressure variations around tracheal intubation | before, during and for 5 minutes after tracheal intubation
  mmHg
Heart rate variations around tracheal intubation | before, during and for 5 minutes after tracheal intubation
  bpm
NOL variation (NOL is an index without unit) around tracheal intubation | before, during and for 5 minutes after tracheal intubation
  Varies from 0 to 100, no unit
Bispectral index (BIS) variation (BIS is an index without unit) around tracheal intubation | before, during and for 5 minutes after tracheal intubation
  Varies from 0 to 100, no unit

CONTACTS AND LOCATIONS:
Locations (1):
- Maisonneuve Rosemont Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No